CLINICAL TRIAL: NCT04692506
Title: A Double-blind, Randomised, Placebo-controlled, Parallel-group Study Evaluating the Safety and Tolerability of Bifidobacterium Longum DSM 32947 Administered to Healthy Volunteers for 28 Days.
Brief Title: Study Evaluating the Safety and Tolerability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioGaia AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CSUB0186
Record Dates: First submitted 2020-12-16; First posted 2020-12-31 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Adouble-blind, randomised, placebo-controlled, parallel-group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study and the allocation of treatments will not be disclosed until clean file has been declared and the database has been locked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose: Sachet with B. longum (Active Comparator): The IP will be self-administered by the subject. Subjects will be asked to consume the IP (1 sachet) once per day, at approximately the same time every day, for 28 days.
  The sachet should be emptied in, and mixed with, a bottle of milk.
  Interventions: Other: Probiotic
- High dose: Sachet with B. longum (Active Comparator): The IP will be self-administered by the subject. Subjects will be asked to consume the IP (1 sachet) once per day, at approximately the same time every day, for 28 days.
  The sachet should be emptied in, and mixed with, a bottle of milk.
  Interventions: Other: Probiotic
- Placebo Sachet (Placebo Comparator): The IP will be self-administered by the subject. Subjects will be asked to consume the IP (1 sachet) once per day, at approximately the same time every day, for 28 days.
  The sachet should be emptied in, and mixed with, a bottle of milk.
  Interventions: Other: Probiotic

INTERVENTIONS:
Other: Probiotic — The study product is probiotic

SUMMARY:
The rationale for the current study is to initially evaluate the safety and tolerability of B. longum strain in healthy volunteers.

DETAILED DESCRIPTION:
The design of the study is based on the aim to study safety and tolerability of B. longum in a limited number of healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Healthy male or female subject aged 18-65 years inclusive.
3. Body Mass Index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2.
4. Clinically normal medical history, physical findings, vital signs, and laboratory values at the time of screening, as judged by the Investigator.
5. Women of child bearing potential (WOCBP) must practice abstinence (only allowed when this is the preferred and usual lifestyle of the subject) or must agree to use a highly effective method of contraception with a failure rate of < 1% to prevent (combined [oestrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, implantable], intrauterine device [IUD]or intrauterine hormone-releasing system [IUS]) from at least 4 weeks prior to dose to 4 weeks after last dose.

Women of non-childbearing potential are defined as pre-menopausal females who are sterilised (tubal ligation or permanent bilateral occlusion of fallopian tubes); or post-menopausal defined as 12 months of amenorrhea (in questionable cases a blood sample with simultaneous detection of follicle stimulating hormone [FSH] 25-140 IE/L is confirmatory).

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IP.
3. Malignancy within the past 5 years with the exception of in situ removal of basal cell carcinoma.
4. Any planned major surgery within the duration of the study.
5. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibodies or HIV.
6. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to Bifidobacterium probiotic treatment.
7. History of, or ongoing GI disorder, including but not limited to irritable bowel syndrome (IBS), constipation, loose stools or excess gas which, in the discretion of the Investigator, may influence the results or the subject's ability to participate in the study.
8. Lactose intolerance (that in the opinion of the Investigator would interfere with the use of yoghurt drinks once daily for 28 days).
9. Regular use of any prescribed or non-prescribed medication including antacids and analgesics within 2 weeks prior to the first administration of IP, at the discretion of the Investigator.
10. Any use of antibiotics (except local treatment, e.g. eye drops) within two weeks prior to the first administration of IP.
11. Planned treatment or treatment with an investigational drug within 3 months prior to Day 1. Subjects consented and screened but not dosed in previous phase I studies are not excluded.
12. Current smokers or users of nicotine products. Irregular use of nicotine (e.g. smoking, snuffing, chewing tobacco) less than three times per week is allowed before screening visit.
13. Positive screen for drugs of abuse or alcohol at screening or on admission to the unit prior to administration of the IP.
14. History of alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
15. Presence or history of drug abuse, as judged by the Investigator.
16. History of, or current use of, anabolic steroids, as judged by the Investigator.
17. Excessive caffeine consumption defined by a daily intake of >5 cups of caffeine
18. Plasma donation within one month of screening or blood donation (or corresponding blood loss) during the three months prior to screening.
19. Investigator considers the subject unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
To evaluate the incidence of treatment emergent adverse events ( safety and tolerability) of B. longum administered to healthy subjects for 28 days. | 28 Days
  The product to be investigated is a probiotic not an investigational medicinal. However, the procedures for monitoring, collecting and reporting of AEs will be the same as for an investigational medicinal product.
  Vital signs, systolic and diastolic blood pressure and pulse will be measured in supine position after 10 minutes of rest. Vital signs will be judged as normal, abnormal, not clinically significant or abnormal, clinically significant.
  Safety laboratory parameters, blood samples for analysis of clinical chemistry and haematology will be analysed by routine analytical methods.
  Urine drug screen analysis will be performed using dip sticks. Urine pregnancy tests will be performed.
  Abnormal values assessed by the Investigator as clinically significant will be reported as AEs. If an abnormal value is associated with corresponding clinical signs or symptoms, the sign/symptom should be reported as the AE.

SECONDARY OUTCOMES:
To evaluate tolerability in terms of gastrointestinal (GI) symptoms during 28 days | 28 Days
  To evaluate gastrointestinal symptoms by using Gastrointestinal Symptom Rating Scale( GSRS) over the last week. The questionnaire will be answered by the subjects at Visits 2 to 5 The GSRS is a disease-specific instrument. The 15 items combine into five symptom clusters: Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation. The reliability and validity of the GSRS are well-documented, and norm values for a general population are available.
  The data collected using the GSRS does not constitute AEs and will not be reported as such but will be reported as numerical results. Accordingly, no causality assessment by the Investigator will be performed for the GSRS questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Rein-Hedin, MD, Principal Investigator — CTC Clinical Trial Consultants AB Dag Hammarskjölds väg 10B SE-752 37 Uppsala, Sweden
Locations (1):
- CTC, Dag Hammarskjölds väg 10B, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No